CLINICAL TRIAL: NCT01069276
Title: Prehospital Transcranial Duplex in Patients With Acute Stroke
Status: Withdrawn | Type: Observational
Why Stopped: Changes in preclinical treatment of stroke patients, no more emergency physician will met this patients
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Patrick Schramm, MD, Johannes Gutenberg University Mainz
Other Study IDs: 837.041.08; 6038 (Registry Identifier: local ethic comitee)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Stroke
Keywords: Stroke; prehospital ultrasound
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with clinical signs of stroke: Patients with clinical signs of stroke
  Interventions: Other: No intervention in this study

INTERVENTIONS:
Other: No intervention in this study — No intervention in this study

SUMMARY:
The aim of the study is to investigate patients with acute stroke prehospital with transcranial duplex ultrasound to detect an infarct of the middle cerebral artery.

DETAILED DESCRIPTION:
The investigation of the patients will be done by an anaesthesiologist who is part of the prehospital medical treatment in Germany. The main question is, wether a non neurologist can detect an infarction of the middle cerebral artery in a short time an lead the patient to the indicated clinic.

ELIGIBILITY:
Inclusion Criteria:

* clinical signs of acute stroke
* possibility of TCD

Exclusion Criteria:

* acute interventions for vital signs required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical signs of acute stroke in the teritorial of the middle cerebral artery
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Prehospital detection of an infarction of the middle cerebral artery in patients with acute stroke | 5 Minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center of the Johannes Gutenberg-University Mainz, Mainz, Germany